CLINICAL TRIAL: NCT00479804
Title: Non-Invasive Determination of Cardiac Output by the Inertgas Rebreathing Method Compared With Magnetic Resonance Tomography
Brief Title: Non-Invasive Determination of Cardiac Output by Inertgas Rebreathing Method
Acronym: NICO
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Dr. Joachim Saur, University Hospital Mannheim
Other Study IDs: 2006-067M-MA
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Cardiac Diseases
Keywords: indication for CMR
MeSH Terms: conditions — Heart Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: inertgas rebreathing — determination of cardiac output by inertgas rebreathing
Device: spirometry — spirometry for testing the ventilatory function
Device: cardiac magnetic resonance imaging (CMR) — CMR examination which delivers the hemodynamic reference parameters

SUMMARY:
The cardiac output (CO) is an important parameter in the diagnosis and therapy of cardiac diseases. The current standard methods for the determination of the CO, however, are either invasive (e.g. right heart catheterization) or technically expendable and expensive (magnetic resonance tomography, MRT). The traditional non-invasive methods of determining the CO by rebreathing of carbon dioxide are easily carried out but suffer from methodical inaccuracies. Therefore the aim of the study at hand was to evaluate a new method for determining the CO by means of the inert gas rebreathing method.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CMR
* Ability of following instructions for rebreathing test

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with indication for CMR
Enrollment: 311 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Saur, Dr., Study Director — 1st Department of Medicine; Jens Kaden, Dr., Study Chair — 1st Deparment of Medicine
Locations (1):
- 1st Department of Medicine, University Hospital Mannheim, Mannheim, Baden-Wurttemberg, Germany